CLINICAL TRIAL: NCT00820677
Title: Innovative Delivery of Newborn Anticipatory Guidance: The Incorporation of Media-Based Learning Into the Primary Care Office.
Brief Title: Newborn Health Information Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: The Commonwealth Fund (Other); Academic Pediatric Association (Industry)
Responsible Party: Heather Paradis, MD, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RSRB00024779
Record Dates: First submitted 2009-01-08; First posted 2009-01-12 (Estimated); Last update posted 2009-12-14 (Estimated); Status verified 2009-01

CONDITIONS: Infant, Newborn

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- DVD/Video (Experimental): Parents of newborns in the experimental group attending their first baby visit will be shown a video about newborn care.
  Interventions: Behavioral: DVD/Video

INTERVENTIONS:
Behavioral: DVD/Video — One DVD or Video will be watched by all parents of newborns enrolled into the experimental group.

SUMMARY:
This is a randomized, controlled trial to test the use of an educational video during the newborn well-child visit. Parents who watch the video during their medical visit will be compared to those parents who receive traditional paper handouts. Measures obtained at baseline and 2-week follow-up include knowledge of infant development, self-efficacy with infant care, and problem-solving skills.

ELIGIBILITY:
Inclusion Criteria:

* Baby's first visit to the pediatric office

Exclusion Criteria:

* Baby > 1 month old
* Parent/Caregiver < 18yrs old
* Inability to understand English
* No access to a working telephone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Knowledge of Infant Development | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Heather A Paradis, MD, Principal Investigator — University of Rochester; Jill S Halterman, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

REFERENCES:
- [Derived] Paradis HA, Conn KM, Gewirtz JR, Halterman JS. Innovative delivery of newborn anticipatory guidance: a randomized, controlled trial incorporating media-based learning into primary care. Acad Pediatr. 2011 Jan-Feb;11(1):27-33. doi: 10.1016/j.acap.2010.12.005. PMID 21272821